CLINICAL TRIAL: NCT01057888
Title: Randomized Controlled Trial of an Automated, Managed Care-based Reminder/Recall System on Improving Rates of Immunization and Preventive Care Visits for Publically Insured Adolescents
Brief Title: Evaluation of Vaccination Reminder/Recall Systems for Adolescent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter G Szilagyi MD MPH, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RSRB00026761
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Immunization Status; Well Child Care Visit
Keywords: Immunization status for:; Tdap; Menactra; HPV (if female); Well child care visit
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Autodialer (Experimental): Autodialer reminder/recall
  Interventions: Other: Autodialer
- Letters (Experimental): Mailed reminder letters
  Interventions: Other: Letters
- Controls (No Intervention): Controls

INTERVENTIONS:
Other: Autodialer — Autodialer telephone calls
  Arms: Autodialer
Other: Letters — Mailed reminder letters
  Arms: Letters

SUMMARY:
The investigators will design and implement a randomized clinical trial to test, on a community-wide level, the effectiveness of managed care based tracking/reminder/recall on improving vaccination coverage among adolescents.

The investigators propose a randomized controlled trial to evaluate the effectiveness of reminder/recall for adolescents: 10,599 adolescents within the managed care organization (MCO) will be randomized into one of three arms: 1) mailed reminders, 2) autodialer telephone messages or 3) standard of care of their practice (no messages from the intervention).

Hypothesis 1: Reminder/recall will increase the receipt of immunizations and preventive services

Hypothesis 2: Telephone (autodialer) reminders will be more effective than mailed reminders

Hypothesis 3: The impact of reminders will be greatest for the most high-risk subgroups which have low baseline immunization rates.

Hypothesis 4: Mailed reminders will be more costly (and less effective) than telephone reminders.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Monroe Plan for Medical Care (managed care organization)
* Patient of a participating practice
* Ages 10.75 to <18 years of age

Exclusion Criteria:

* Member of the Monroe Plan for Medical care for less than 6 months
* ICD-9 diagnosis of 999.4 for anaphylactic reaction to a vaccine or its components.
* Encephalopathy within 7 days of a previous dose of a pertussis containing vaccine not attributable to another identifiable cause
* Guillain-Barre- ICD-9 code is 357.0

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10599 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Szilagyi, MD, MPH, Principal Investigator — University of Rochester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From the managed care plan's dataset of practices, we selected all primary care practices that served >30 adolescents covered by the managed care plan in December 2009. The target population was all adolescents ages 10.5 through 17 years enrolled in Monroe Plan on December 31st 2009 with a primary care provider in a participating practice.
Pre-assignment Details: One individual was assessed for randomization, was found to have a previous case of anaphylaxis and was not randomized.
Groups:
- Autodialer: Autodialer reminder/recall
  Autodialer : Autodialer telephone calls
- Controls: Controls
  Received standard of care provided by practice
- Letters: Mailed reminder letters
  Letters : Mailed reminder letters
Period: Overall Study
Arm/Group | Autodialer | Controls | Letters
Started | 2504 | 2406 | 2494
Completed | 2504 | 2406 | 2494
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autodialer | Controls | Letters | Total
Number analyzed (Participants) | 1423 | 1296 | 1396 | 4115
Age, Categorical [Number; unit: participants]
  <=18 years | 1,423 | 1,296 | 1,396 | 4115
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.0) | 14.5 (2.0) | 14.4 (2.0) | 14.4 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 699 | 656 | 682 | 2037
  Male | 724 | 640 | 714 | 2078

OUTCOME MEASURES:

1. Primary Outcome: Fully Vaccinated (Tdap, Menactra and 3 Doses of HPV (if Female))
Time Frame: 12 months
Population: Individuals were randomized to one of 3 groups (letter reminders, telephone reminders or control). Individuals with a wrong/missing telephone number or a wrong address were excluded from the analyses. This left 1,396 in the letter reminder group, 1,423 in the telephone reminder group and 1,296 in the control group.
Measure: Number; unit: participants
Groups:
- Letter Reminder: Received mailed reminders from the managed-care organization for recommended vaccinations
- Telephone Reminder: Received telephone reminders (through an autodialer)from the managed-care organization for recommended vaccinations
- Control: Received no reminders from the managed care organization.
Arm/Group | Letter Reminder | Telephone Reminder | Control
Number analyzed (Participants) | 1396 | 1423 | 1296
participants | 143 | 160 | 100
Statistical Analysis 1: Comparison: Telephone Reminder vs Control; The null hypothesis is that there is no difference in total immunization status between the control group and the group receiving telephone (autodialer) reminders. This was analyzed using a clustered, stratified Cox model; Test type: Superiority or Other; p < 0.05, Regression, Cox; It is a robust, clustered stratified Cox regression model; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [1.0 to 1.7] — The control group serves as the denominator. The telephone reminder group serves as the numerator
Statistical Analysis 2: Comparison: Letter Reminder vs Control; Test type: Superiority or Other; p < 0.01, Regression, Cox; We used a robust, clustered, stratified Cox regression model; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [1.3 to 2.1] — The control group represents the denominator. The letter reminder group represents the numerator
Statistical Analysis 3: Comparison: Letter Reminder vs Telephone Reminder; The null hypothesis was that there is no difference in the percentage of fully vaccinated adolescents between the mailed reminder versus the telephone reminder arms; Test type: Superiority or Other; p = 0.075, Regression, Cox; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [1.0 to 1.6] — The mail reminder arm represents the numerator and the telephone reminder arm represents the denominator

2. Primary Outcome: Well Child Care Status
Description: Received recommended well child care visit
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Letter Reminder | Telephone Reminder | Control
Number analyzed (Participants) | 1396 | 1423 | 1296
participants | 908 | 892 | 768
Statistical Analysis 1: Comparison: Letter Reminder vs Control; The null hypothesis was that a difference in well child care rates among adolescents whose families received a mailed reminder compared to the control group; Test type: Superiority or Other; p < 0.01, Regression, Cox; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [1.1 to 1.3] — The control group represents the denominator and the mailed reminder group represents the numerator
Statistical Analysis 2: Comparison: Telephone Reminder vs Control; The null hypothesis is the the well child care rates of adolescents in the telephone reminder group would not differ from those of the control group; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [1.0 to 1.3] — The control group represents the denominator and the telephone reminder group represents the numerator
Statistical Analysis 3: Comparison: Letter Reminder vs Telephone Reminder; The null hypothesis was that there would be no difference in the well child care rate among adolescents in the mailed reminder arm versus adolescents in the telephone reminder arm of the intervention; Test type: Superiority or Other; p = 0.234, Regression, Cox; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [1.0 to 1.2] — The mail reminder arm represents the numerator and the telephone reminder arm represents the denominator

ADVERSE EVENTS:
Time Frame: N/A- reviewed claims data
Arm/Group | Mailed Reminders and Letter Reminders
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No